CLINICAL TRIAL: NCT06958042
Title: Investigation of the Prevalence of Lower Urinary Tract Symptoms and the Level of Knowledge About Pelvic Floor Health in Individuals With Chronic Obstructive Pulmonary Disease
Brief Title: The Prevalence of Lower Urinary Tract Symptoms in Individuals With Chronic Obstructive Pulmonary Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Gamze Kurt, Assos. Prof., Kutahya Health Sciences University
Other Study IDs: COPD_INCONTINENCE
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Incontinance; Pelvic floor muscle
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire and Physical Exam — - St George Respiratory Questionnaire (SGRQ): The SGRQ developed by Jones (2000), which is used specifically for respiratory diseases, consists of 50 questions. In the questionnaire, there are three categories in which symptom, activity and the effect of the disease on quality of life are questioned and each category is evaluated within itself and there is an evaluation scale between 0-100 points. In the evaluation, high scores indicate an inadequate and low quality of life.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic lung disease characterized by airflow limitations and respiratory symptoms due to structural changes in the airways. Common symptoms include dyspnea, chronic cough, and increased sputum production. Respiratory diseases are a risk factor for lower urinary tract symptoms, which can lead to leakage if pelvic floor muscles are weak. Lower urinary tract symptoms are classified into storage, emptying, and post-emptying groups. Current literature on urinary incontinence in COPD patients is limited, and there is a need for further research on the presence and effects of lower urinary system symptoms in individuals with COPD and the level of pelvic floor health knowledge.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is defined as a chronic lung disease characterized by progressive airflow limitation and chronic respiratory symptoms due to structural changes in the airways. Dyspnea (shortness of breath), chronic cough, and increased sputum production are the most common symptoms in individuals with COPD. Respiratory diseases are considered a risk factor for lower urinary tract symptoms due to cough and shortness of breath. Severe coughing and shortness of breath increase intra-abdominal pressure and stress on the bladder. These conditions can lead to leakage if the pelvic floor muscles are weak. In addition, regular coughing can further weaken the ligaments in the pelvic floor, causing symptoms.

Lower urinary tract symptoms is a general term covering various functional disorders of the bladder, pelvic floor, or specific pathologies. The International Continence Society classifies lower urinary tract symptoms in three main groups: storage (increased/decreased urination, urinary incontinence, nocturia, overactive bladder), emptying (delayed urination, painful urination, intermittent urination), and post-emptying (feeling of not being able to empty the bladder completely, repeated urge to urinate, urinary tract infections). When the current literature was examined, it was observed that there are studies on the presence of urinary incontinence in patients with chronic respiratory disease, but there are limited studies investigating the presence and effects of lower urinary system symptoms in individuals with COPD in general and investigating the level of pelvic floor health knowledge. In this context, our study is unique and may contribute to future rehabilitation studies in this field.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD (according to GOLD criteria)
* Being clinically stable
* Volunteering to participate in the study

Exclusion Criteria:

* Having perception and cognitive problems
* Having a diagnosis of unstable COPD

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients who agreed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Incontinence Quality of Life Scale (IQOL) | Enrolllment
  The Turkish validity and reliability studies of the scale developed by Patrick et al. (1999) to determine the quality of life of patients with urinary incontinence were conducted by Özerdoğan et al. There are 22 questions in the scale and each question is evaluated with a Likert-type scale divided into five categories (1: very much, 2: quite, 3: moderately, 4: a little, 5: not at all). IQOL has three sub-dimensions: limiting behaviour, psychological impact and limiting social life. The total score of the scale ranges from 0-100 and it is concluded that the higher the score, the better the quality of life level.
St George Respiratory Questionnaire (SGRQ) | Enrollment
  Quality of life will be evaluated using the SGRQ, which includes symptoms, activity, and impact domains.
  Scores range from 0 to 100, with higher scores indicating poorer quality of life.

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | Enrollment
  The ICIQ-SF was developed by the International Consultation on Incontinence to assess the frequency, severity and impact of incontinence. The scale consists of four dimensions. The first dimension assesses how often incontinence occurs, the second dimension assesses the amount of incontinence, the third dimension assesses the effect of incontinence on daily life and the last dimension assesses the conditions that cause incontinence. The first three dimensions are included in the scoring and the fourth dimension is used to determine the type of incontinence. The total score of the scale varies between 0-21 and an increase in score indicates an increase in severity.
International Consultation on Incontinence Questionnaire-Male Lower Urinary System Symptoms (ICIQ-MLUTS) | Enrollment
  Turkish validity and reliability studies of the ICIQ-MLUTS scale developed by the International Consultation on Incontinence to evaluate lower urinary system symptoms in male individuals were conducted by Mertoğlu et al. The scale consists of 13 items in total. 5 items question voiding symptoms, 6 items question storage symptoms, frequent daytime urination and number of nighttime urination. The items in the storage and voiding subsections question the presence and severity of the symptom and rate it according to a Likert scale (0: Never, 1: Rarely, 2: Occasionally, 3: Mostly, 4: Always). The voiding symptom score of the scale is 0-20 and the storage symptom score is 0-24.
International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) | Enrollment
  The Incontinence Questionnaire - Female Lower Urinary Tract Symptoms Long Form (ICIQ-FLUTS-LF) was divided into 6 subgroups of symptom measurements, which were storage, voiding, incontinence, bladder pain, post-micturition, and ability to stop voiding. Each severity item is rated from 0 to 4, and each bothersome item from 0 to 10. The total severity score ranges from 0 to 20, and the total bothersome score ranges from 0 to 50. Higher scores indicate worse outcomes.

OTHER OUTCOMES:
Pelvic Floor Health Knowledge Test | Enrollment
  according to the subscales of this test: pelvic floor function/dysfunction (8 items), risk factors of pelvic floor dysfunctions (18 items), and diagnosis and treatment of 11 items. All items were created simply and understandably with three response categories: "yes," "no," and "I do not know." A dichotomous system was used for scoring: "1" point for the items that were answered correctly and "0" points for the items that were answered incorrectly or unknown.
Prolapse and Incontinence Knowledge Questionnaire | Enrollment
  The participants read and indicated their agreement levels (agree, disagree, do not know) with 24 items (12 items for each subscale) in this knowledge scale. Each item has a correct response, and the participants were given a "1" point if they have marked that response. Incorrect, missing, or "don't know" answers were scored as "0" points. Scores of subscales (0-12 points), and the overall scale (0-24 points) were calculated, and higher scores indicated a higher level of knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Helath Sciences University- Health Sciences Faculty, Kütahya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided